CLINICAL TRIAL: NCT01608100
Title: Design Validation Protocol for the Evaluation of ARCHITECT STAT High Sensitive Troponin I Assay
Brief Title: Evaluation of a New Cardiac Biomarker Assay
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Diagnostics Division (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7B5-02-10A01-03
Record Dates: First submitted 2012-05-21; First posted 2012-05-30 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-01

CONDITIONS: Acute Coronary Syndrome; Acute Myocardial Infarction
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARCHITECT STAT High Sensitive Troponin I Assay testing (Experimental): All subjects will have their blood tested by the investigational ARCHITECT STAT High SensitiveTroponin I assay.
  Interventions: Device: ARCHITECT STAT High Sensitive Troponin I Assay

INTERVENTIONS:
Device: ARCHITECT STAT High Sensitive Troponin I Assay — Test blood samples from the ARCHITECT STAT High Sensitive Troponin I Assay. Results obtained will be used to assess the prognosis of subjects for risk of ACM/MACE in the timeframes (30 days and 90 days) after the Emergency Department visit.
  Troponin results will be compared to documented ACM/MACE events at the 30 day and 90 day time points after Emergency Department visit.

SUMMARY:
The objective of the study is to evaluate the performance and intended use of a new cardiac biomarker test, Troponin I, in an intended use population. Blood specimens will be tested using the new investigational test that detects the level of Troponin I. Results will be compared to the diagnosis of whether or not an acute myocardial infarction (MI) occurred.

DETAILED DESCRIPTION:
The purpose of the cardiac biomarker Troponin I is to aid in the diagnosis of myocardial infarction.The assay is also intended to assist in the prognosis relative risk to all cause mortality (ACM) and major adverse cardiac events (MACE) consisting of myocardial infarction, revascularization, and cardiac death in patients who present with symptoms suggestive of acute coronary syndrome (ACS) without a diagnosis of myocardial infarction.

All specimens were collected under a separate specimen collection protocol (Protocol No, 7B5-02-09A01-01: Clinical Specimen Procurement for Biomarker Evaluation of Suspected ACS). The specimens that will be tested include approximately 8300 specimens collected from 1101 subjects presenting to Emergency Departments with signs and symptoms of Acute Coronary Syndrome and will be provided to the clinical sites performing investigational Troponin I testing.

ELIGIBILITY:
Inclusion Criteria:

* presenting to the Emergency Department with symptoms consistent with or suggestive of Acute Coronary Syndrome (ACS) defined as at least 5 minutes of chest pain (or symptoms consistent with myocardial ischemia) up to 6 hours prior to initial evaluation.
* an Electrocardiogram (ECG) result within 2 hours of presentation for observation of Acute Coronary Syndrome (ACS).
* greater than 18 years of age.
* not known to be pregnant.
* agreement to the follow-up required by the study.

Exclusion Criteria:

* prior participation in this study.
* require dialysis for end stage renal disease.
* history of a previous heart transplant.
* coexisting disorder associated with limited life expectancy.
* currently participating in another investigational device or drug study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1101 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred S Apple, PhD, Principal Investigator — Hennepin Healthcare Research Institute; Frank Peacock, MD, Study Chair
Locations (12):
- United States (12):
  - Chandler Regional Medical Center, Chandler, Arizona
  - Stanford University School of Emergency Medicine, Palo Alto, California
  - Nationwide Laboratory Services, Fort Lauderdale, Florida
  - John T Mather Memorial Hospital, Port Jefferson, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Pennsylvania State University- Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hospital Physicians in Clinical Research, Austin, Texas
  - Hospital Physicians in Clinical Research, Bryan, Texas
  - Dept of Emergency Medicine University of Virginia, Charlottesville, Virginia
  - St Joseph Hospital, Bellingham, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- ARCHITECT STAT High Sensitive Troponin I Assay Testing: All subjects will have their blood tested by the investigational Troponin I assay.
  ARCHITECT STAT High Sensitive Troponin I Assay: Test blood samples from the ARCHITECT STAT High Sensitive Troponin I Assay.
  Results obtained will be used to assess the prognosis of subjects for risk of ACM/MACE in the time frames (30 days and 90 days) after the Emergency Department visit.
  Troponin results will be compared to documented ACM/MACE events at the 30 day and 90 day time points after Emergency Department visit.
Period: Overall Study
Arm/Group | ARCHITECT STAT High Sensitive Troponin I Assay Testing
Started | 1101
Completed | 1101
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- ARCHITECT STAT High Sensitive Troponin I Assay Testing: All subjects will have their blood tested by the investigational ARCHITECT STAT High Sensitive Troponin I assay. Specimens were collected at 11 emergency departments from 1,101 subjects presenting to the emergency department with symptoms consistent with acute coronary syndrome (ACS). All subject diagnoses were adjudicated by three board certified cardiologists according to current standard of care.
Arm/Group | ARCHITECT STAT High Sensitive Troponin I Assay Testing
Number analyzed (Participants) | 1101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 746
  >=65 years | 355
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 482
  Male | 619
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 300
  White | 692
  Hispanic | 62
  Asian | 18
  Other | 29
Observed Myocardial Infarction Prevalence [Number; unit: participants]
  Number Participants with Myocardial Infarction | 130
  Number Participants without Myocardial Infarction | 971

OUTCOME MEASURES:

1. Primary Outcome: Clinical Performance - Area Under the Curve
Description: The ARCHITECT STAT High Sensitive Troponin-I assay clinical performance was evaluated by calculating the Area Under the Curve (AUC). The Area Under the Curve that was assessed, is used to determine the optimum clinical sensitivity and specificity for the ARCHITECT STAT High Sensitive Troponin-I assay. The ARCHITECT STAT High Sensitive Troponin-I assay results were generated from subject's specimens collected at three collection time points in three tube types (K2 EDTA, Lithium Heparin Separator and Serum Separator).
Time Frame: Troponin value from three collection time points (0-2 hours, >2 and up to 4 hours, >4 hours and up to 9 hours) from subject presentation to the emergency department
Population: The number of subjects for analysis was determined by the number of subjects with at least one collection time point in the respective tube type (K2 EDTA, Lithium Heparin Separator, Serum Separator). Not all time points or collection tube types were able to be collected for all subjects.
Measure: Number (95% Confidence Interval); unit: Probability
Groups:
- Area Under the Curve in K2 EDTA: Area Under the Curve for the ARCHITECT High Sensitive Troponin I was evaluated using K2 EDTA tube type for 3 collection time points. The results were calculated using the overall 99th percentile cutoff (26.2 pg/mL).
- Area Under the Curve in Lithium Heparin Separator: Area Under the Curve for the ARCHITECT High Sensitive Troponin I was evaluated using Lithium Heparin tube type for 3 collection time points. The results were calculated using the overall 99th percentile cutoff (26.2 pg/mL).
- Area Under the Curve in Serum Separator: Area Under the Curve for the ARCHITECT High Sensitive Troponin I was evaluated using Serum tube type for 3 collection time points. The results were calculated using the overall 99th percentile cutoff (26.2 pg/mL).
Arm/Group | Area Under the Curve in K2 EDTA | Area Under the Curve in Lithium Heparin Separator | Area Under the Curve in Serum Separator
Number analyzed (Participants) | 1066 | 1088 | 1029
Probability
  Area Under the Curve: 0-2 hours | 0.9326 [0.9048 to 0.9604] | 0.9197 [0.8914 to 0.9480] | 0.9412 [0.9102 to 0.9722]
  Area Under the Curve: 2-4 hours | 0.9431 [0.9081 to 0.9782] | 0.9349 [0.8986 to 0.9712] | 0.9419 [0.9041 to 0.9796]
  Area Under the Curve: 4-9 hours | 0.9503 [0.9419 to 0.9857] | 0.9498 [0.9190 to 0.9805] | 0.9449 [0.9046 to 0.9852]
Statistical Analysis 1: Comparison: Area Under the Curve in K2 EDTA; Time point: 0-2 hours; Test type: Superiority or Other; Area Under the Curve = 0.9326, 95% CI 2-sided [0.9048 to 0.9604]
Statistical Analysis 2: Comparison: Area Under the Curve in K2 EDTA; Time point: 2-4 hours; Test type: Superiority or Other; Area Under the Curve = 0.9431, 95% CI 2-sided [0.9081 to 0.9782]
Statistical Analysis 3: Comparison: Area Under the Curve in K2 EDTA; Time point: 4-9 hours; Test type: Superiority or Other; Area Under the Curve = 0.9503, 95% CI 2-sided [0.9419 to 0.9857]
Statistical Analysis 4: Comparison: Area Under the Curve in Lithium Heparin Separator; Time point: 0-2 hours; Test type: Superiority or Other; Area Under the Curve = 0.9197, 95% CI 2-sided [0.8914 to 0.9480]
Statistical Analysis 5: Comparison: Area Under the Curve in Lithium Heparin Separator; Time point: 2-4 hours; Test type: Superiority or Other; Area Under the Curve = 0.9349, 95% CI 2-sided [0.8986 to 0.9712]
Statistical Analysis 6: Comparison: Area Under the Curve in Lithium Heparin Separator; Time point: 4-9 hours; Test type: Superiority or Other; Area Under the Curve = 0.9498, 95% CI 2-sided [0.9190 to 0.9805]
Statistical Analysis 7: Comparison: Area Under the Curve in Serum Separator; Time point: 0-2 hours; Test type: Superiority or Other; Area Under the Curve = 0.9412, 95% CI 2-sided [0.9102 to 0.9722]
Statistical Analysis 8: Comparison: Area Under the Curve in Serum Separator; Time point: 2-4 hours; Test type: Superiority or Other; Area Under the Curve = 0.9419, 95% CI 2-sided [0.9041 to 0.9796]
Statistical Analysis 9: Comparison: Area Under the Curve in Serum Separator; Time point: 4-9 hours; Test type: Superiority or Other; Area Under the Curve = 0.9449, 95% CI 2-sided [0.9046 to 0.9852]

2. Secondary Outcome: Prognosis
Description: Specimens were collected at 11 EDs from 1,101 subjects presenting to the ED with symptoms consistent with ACS. All subject diagnoses were adjudicated by three board certified cardiologists according to current standard of care. ARCHITECT STAT High Sensitive Troponin I results were generated from subject specimens and evaluated for use as an aid in the assessment of prognosis. Analyses used the first available troponin result from multiple serial draw time points. Subjects were assessed for risk of all cause mortality (ACM) and major adverse cardiac event (MACE) at 30 day and 90 day time points after ED discharge. MACE consisted of myocardial infarction, urgent revascularization, and cardiac death. Subjects were followed-up for subsequent events by medical record review and/or subject/caregiver contact. Any ACM and MACE that occurred during the ED visit and on the same day as ED discharge were not included in the analyses.
Time Frame: 30-day and 90-day follow-up
Population: 30 Day and 90-day prognosis (Kaplan Meier analysis) and Hazard ratios (Cox regression) for the overall 99th percentile cutoff (26.2 pg/mL) are summarized. *Censored is defined as the subject has not experienced ACM/MACE at the indicated follow-up time point.
Measure: Number; unit: participants
Groups:
- 30-day Prognosis for K2 EDTA Tube Type; 30-day Prognosis for Lithium Heparin Separator Tube Type; 30-day Prognosis for Serum Separator Tube Type: The 30-day prognosis (Kaplan-Meier analysis) and hazard ratios (Cox regression) for the overall 99th percentile cutoff (26.2 pg/mL) were calculated.
- 90-day Prognosis for K2 EDTA Tube Type; 90-day Prognosis for Lithium Heparin Separator Tube Type; 90-day Prognosis for Serum Separator Tube Type: The 90-day prognosis (Kaplan-Meier analysis) and hazard ratios (Cox regression) for the overall 99th percentile cutoff (26.2 pg/mL) were calculated.
Arm/Group | 30-day Prognosis for K2 EDTA Tube Type | 90-day Prognosis for K2 EDTA Tube Type | 30-day Prognosis for Lithium Heparin Separator Tube Type | 90-day Prognosis for Lithium Heparin Separator Tube Type | 30-day Prognosis for Serum Separator Tube Type | 90-day Prognosis for Serum Separator Tube Type
Number analyzed (Participants) | 1064 | 1064 | 1085 | 1085 | 1027 | 1027
participants
  MACE/ACM with Troponin value </= cutoff | 19 | 30 | 17 | 30 | 17 | 29
  No MACE/ACM (*Censored) with TnI value </= cutoff | 802 | 791 | 803 | 790 | 796 | 784
  MACE/ACM with Troponin value > cutoff | 17 | 31 | 19 | 34 | 13 | 26
  No MACE/ACM (*Censored) with TnI value > cutoff | 226 | 212 | 246 | 231 | 201 | 188
Statistical Analysis 1: Comparison: 30-day Prognosis for K2 EDTA Tube Type; Kaplan-Meier; Test type: Superiority or Other; p = 0.0004, Log Rank; Proportion Percentage = 7.00 — Proportion percentage for subjects with ARCHITECT Troponin value greater than the cutoff
Statistical Analysis 2: Comparison: 30-day Prognosis for K2 EDTA Tube Type; Kaplan-Meier; Test type: Superiority or Other; p = 0.0004, Log Rank; Proportion Percentage = 2.31 — Proportion percentage for subjects with ARCHITECT Troponin value less than or equal to the cutoff
Statistical Analysis 3: Comparison: 30-day Prognosis for K2 EDTA Tube Type; Hazard Ratio; Test type: Superiority or Other; p = 0.0011, Regression, Cox — Likelihood Ratio; Hazard Ratio (HR) = 3.09, 95% CI 2-sided [1.59 to 5.95]
Statistical Analysis 4: Comparison: 90-day Prognosis for K2 EDTA Tube Type; Kaplan-Meier; Test type: Superiority or Other; p < 0.0001, Log Rank; Proportion Percentage = 12.76 — Proportion percentage for subjects with ARCHITECT Troponin value greater than the cutoff
Statistical Analysis 5: Comparison: 90-day Prognosis for K2 EDTA Tube Type; Kaplan-Meier; Test type: Superiority or Other; p < 0.0001, Log Rank; Proportion Percentage = 3.65 — Proportion percentage for subjects with ARCHITECT Troponin value less than or equal to the cutoff
Statistical Analysis 6: Comparison: 90-day Prognosis for K2 EDTA Tube Type; Hazard Ratio; Test type: Superiority or Other; p < 0.0001, Regression, Cox — Likelihood Ratio; Hazard Ratio (HR) = 3.65, 95% CI 2-sided [2.21 to 6.05]
Statistical Analysis 7: Comparison: 30-day Prognosis for Lithium Heparin Separator Tube Type; Kaplan-Meier; Test type: Superiority or Other; p < 0.0001, Log Rank; Proportion Percentage = 7.17 — Proportion percentage for subjects with ARCHITECT Troponin value greater than the cutoff
Statistical Analysis 8: Comparison: 30-day Prognosis for Lithium Heparin Separator Tube Type; Kaplan-Meier; Test type: Superiority or Other; p < 0.0001, Log Rank; Proportion Percentage = 2.07 — Proportion percentage for subjects with ARCHITECT Troponin value less than or equal to the cutoff
Statistical Analysis 9: Comparison: 30-day Prognosis for Lithium Heparin Separator Tube Type; Hazard Ratio; Test type: Superiority or Other; p = 0.0002, Regression, Cox — Likelihood Ratio; Hazard Ratio (HR) = 3.54, 95% CI 2-sided [1.84 to 6.87]
Statistical Analysis 10: Comparison: 90-day Prognosis for Lithium Heparin Separator Tube Type; Kaplan-Meier; Test type: Superiority or Other; p < 0.0001, Log Rank; Proportion Percentage = 12.83 — Proportion percentage for subjects with ARCHITECT Troponin value greater than the cutoff
Statistical Analysis 11: Comparison: 90-day Prognosis for Lithium Heparin Separator Tube Type; Kaplan-Meier; Test type: Superiority or Other; p < 0.0001, Log Rank; Proportion Percentage = 3.66 — Proportion percentage for subjects with ARCHITECT Troponin value less than or equal to the cutoff
Statistical Analysis 12: Comparison: 90-day Prognosis for Lithium Heparin Separator Tube Type; Hazard Ratio; Test type: Superiority or Other; p < 0.0001, Regression, Cox — Likelihood Ratio; Hazard Ratio (HR) = 3.68, 95% CI 2-sided [2.25 to 6.05]
Statistical Analysis 13: Comparison: 30-day Prognosis for Serum Separator Tube Type; Kaplan-Meier; Test type: Superiority or Other; p = 0.0020, Log Rank; Proportion Percentage = 6.07 — Proportion percentage for subjects with ARCHITECT Troponin value greater than the cutoff
Statistical Analysis 14: Comparison: 30-day Prognosis for Serum Separator Tube Type; Kaplan-Meier; Test type: Superiority or Other; p = 0.0020, Log Rank; Proportion Percentage = 2.09 — Proportion percentage for subjects with ARCHITECT Troponin value less than or equal to the cutoff
Statistical Analysis 15: Comparison: 30-day Prognosis for Serum Separator Tube Type; Hazard Ratio; Test type: Superiority or Other; p = 0.0050, Regression, Cox — Likelihood Ratio; Hazard Ratio (HR) = 2.95, 95% CI 2-sided [1.41 to 6.05]
Statistical Analysis 16: Comparison: 90-day Prognosis for Serum Separator Tube Type; Kaplan-Meier; Test type: Superiority or Other; p < 0.0001, Log Rank; Proportion Percentage = 12.15 — Proportion percentage for subjects with ARCHITECT Troponin value greater than the cutoff
Statistical Analysis 17: Comparison: 90-day Prognosis for Serum Separator Tube Type; Kaplan-Meier; Test type: Superiority or Other; p < 0.0001, Log Rank; Proportion Percentage = 3.57 — Proportion percentage for subjects with ARCHITECT Troponin value less than or equal to the cutoff
Statistical Analysis 18: Comparison: 90-day Prognosis for Serum Separator Tube Type; Hazard Ratio; Test type: Superiority or Other; p < 0.0001, Regression, Cox — Likelihood Ratio; Hazard Ratio (HR) = 3.55, 95% CI 2-sided [2.08 to 6.03]

3. Primary Outcome: Clinical Performance- Sensitivity
Description: The ARCHITECT STAT High Sensitive Troponin-I assay clinical performance was evaluated by calculating Sensitivity. The ARCHITECT STAT High Sensitive Troponin-I assay results were generated from subject's specimens collected at three collection time points in three tube types (K2 EDTA, Lithium Heparin Separator and Serum Separator).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage MI withTnI >cutoff vs all MI
Groups:
- Sensitivity in K2 EDTA: Sensitivity for the ARCHITECT High Sensitive Troponin I was evaluated using K2 EDTA tube type for 3 collection time points. The results were calculated using the overall 99th percentile cutoff (26.2 pg/mL).
- Sensitivity in Lithium Heparin Separator: Sensitivity for the ARCHITECT High Sensitive Troponin I was evaluated using Lithium Heparin tube type for 3 collection time points. The results were calculated using the overall (99th percentile cutoff 26.2 pg/mL).
- Sensitivity in Serum Separator: Sensitivity for the ARCHITECT High Sensitive Troponin I was evaluated using Serum tube type for 3 collection time points. The results were calculated using the overall 99th percentile cutoff (26.2 pg/mL).
Arm/Group | Sensitivity in K2 EDTA | Sensitivity in Lithium Heparin Separator | Sensitivity in Serum Separator
Number analyzed (Participants) | 1066 | 1088 | 1029
percentage MI withTnI >cutoff vs all MI
  % Sensitivity: 0-2 hours | 84.44 [75.28 to 91.23] | 85.26 [76.51 to 91.70] | 87.32 [77.30 to 94.04]
  % Sensitivity: 2-4 hours | 92.21 [83.81 to 97.09] | 91.86 [83.95 to 96.66] | 92.00 [83.40 to 97.01]
  % Sensitivity: 4-9 hours | 93.90 [86.34 to 97.99] | 94.95 [88.61 to 98.34] | 93.15 [84.74 to 97.74]
Statistical Analysis 1: Comparison: Sensitivity in K2 EDTA; Time point: 0-2 hours; Test type: Superiority or Other; Percent Sensitivity = 84.44, 95% CI 2-sided [75.28 to 91.23]
Statistical Analysis 2: Comparison: Sensitivity in K2 EDTA; Time point: 2-4 hours; Test type: Superiority or Other; Percent Sensitivity = 92.21, 83.81% CI 2-sided [83.81 to 97.09]
Statistical Analysis 3: Comparison: Sensitivity in K2 EDTA; Time point: 4-9 hours; Test type: Superiority or Other; Percent Sensitivity = 93.90, 95% CI 2-sided [86.34 to 97.99]
Statistical Analysis 4: Comparison: Sensitivity in Lithium Heparin Separator; Time point: 0-2 hours; Test type: Superiority or Other; Percent Sensitivity = 85.26, 95% CI 2-sided [76.51 to 91.70]
Statistical Analysis 5: Comparison: Sensitivity in Lithium Heparin Separator; Time point: 2-4 hours; Test type: Superiority or Other; Percent Sensitivity = 91.86, 95% CI 2-sided [83.95 to 96.66]
Statistical Analysis 6: Comparison: Sensitivity in Lithium Heparin Separator; Time point: 4-9 hours; Test type: Superiority or Other; Percent Sensitivity = 94.95, 95% CI 2-sided [88.61 to 98.34]
Statistical Analysis 7: Comparison: Sensitivity in Serum Separator; Time point: 0-2 hours; Test type: Superiority or Other; Percent Sensitivity = 87.32, 95% CI 2-sided [77.30 to 94.04]
Statistical Analysis 8: Comparison: Sensitivity in Serum Separator; Time point: 2-4 hours; Test type: Superiority or Other; Percent Sensitivity = 92.00, 95% CI 2-sided [83.40 to 97.01]
Statistical Analysis 9: Comparison: Sensitivity in Serum Separator; Time point: 4-9 hours; Test type: Superiority or Other; Percent Sensitivity = 93.15, 95% CI 2-sided [84.74 to 97.74]

4. Primary Outcome: Clinical Performance- Specificity
Description: The ARCHITECT STAT High Sensitive Troponin-I assay clinical performance was evaluated by calculating Specificity. The ARCHITECT STAT High Sensitive Troponin-I assay results were generated from subject's specimens collected at three collection time points in three tube types (K2 EDTA, Lithium Heparin Separator and Serum Separator).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % nonMI with TnI </= cutoff vs all nonMI
Groups:
- Specificity in K2 EDTA: Specificity for the ARCHITECT High Sensitive Troponin I was evaluated using K2 EDTA tube type for 3 collection time points. The results were calculated using the overall (99th percentile cutoff 26.2 pg/mL).
- Specificity in Lithium Heparin Separator: Specificity for the ARCHITECT High Sensitive Troponin I was evaluated using Lithium Heparin tube type for 3 collection time points. The results were calculated using the overall (99th percentile cutoff 26.2 pg/mL).
- Specificity in Serum Separator: Specificity for the ARCHITECT High Sensitive Troponin I was evaluated using Serum tube type for 3 collection time points. The results were calculated using the overall (99th percentile cutoff 26.2 pg/mL).
Arm/Group | Specificity in K2 EDTA | Specificity in Lithium Heparin Separator | Specificity in Serum Separator
Number analyzed (Participants) | 1066 | 1088 | 1029
% nonMI with TnI </= cutoff vs all nonMI
  % Specificity: 0-2 hours | 85.73 [83.18 to 88.03] | 83.76 [81.12 to 86.17] | 86.35 [83.79 to 88.63]
  % Specificity: 2-4 hours | 85.20 [82.66 to 87.50] | 83.72 [81.09 to 86.11] | 85.81 [83.31 to 88.07]
  % Specificity: 4-9 hours | 82.82 [79.99 to 85.40] | 80.72 [77.82 to 83.39] | 84.05 [81.31 to 86.54]
Statistical Analysis 1: Comparison: Specificity in K2 EDTA; Time point: 0-2 hours; Test type: Superiority or Other; Percent Specificity = 85.73, 95% CI 2-sided [83.18 to 88.03]
Statistical Analysis 2: Comparison: Specificity in K2 EDTA; Time point: 2-4 hours; Test type: Superiority or Other; Percent Specificity = 85.20, 95% CI 2-sided [82.66 to 87.50]
Statistical Analysis 3: Comparison: Specificity in K2 EDTA; Time point: 4-9 hours; Test type: Superiority or Other; Percent Specificity = 82.82, 95% CI 2-sided [79.99 to 85.40]
Statistical Analysis 4: Comparison: Specificity in Lithium Heparin Separator; Time point: 0-2 hours; Test type: Superiority or Other; Percent Specificity = 83.76, 95% CI 2-sided [81.12 to 86.17]
Statistical Analysis 5: Comparison: Specificity in Lithium Heparin Separator; Time point: 2-4 hours; Test type: Superiority or Other; Percent Specificity = 83.72, 95% CI 2-sided [81.09 to 86.11]
Statistical Analysis 6: Comparison: Specificity in Lithium Heparin Separator; Time point: 4-9 hours; Test type: Superiority or Other; Percent Specificity = 80.72, 95% CI 2-sided [77.82 to 83.39]
Statistical Analysis 7: Comparison: Specificity in Serum Separator; Time point: 0-2 hours; Test type: Superiority or Other; Percent Specificity = 86.35, 95% CI 2-sided [83.79 to 88.63]
Statistical Analysis 8: Comparison: Specificity in Serum Separator; Time point: 2-4 hours; Test type: Superiority or Other; Percent Specificity = 85.81, 95% CI 2-sided [83.31 to 88.07]
Statistical Analysis 9: Comparison: Specificity in Serum Separator; Time point: 4-9 hours; Test type: Superiority or Other; Percent Specificity = 84.05, 95% CI 2-sided [81.31 to 86.54]

5. Primary Outcome: Clinical Performance- Negative Predictive Value (NPV)
Description: The ARCHITECT STAT High Sensitive Troponin-I assay clinical performance was evaluated by calculating Negative Predictive Value. The ARCHITECT STAT High Sensitive Troponin-I assay results were generated from subject's specimens collected at three collection time points in three tube types (K2 EDTA, Lithium Heparin Separator and Serum Separator).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: %nonMI,TnI</=cutoff vs all TnI</=cutoff
Groups:
- Negative Predictive Value in K2 EDTA: Negative Predictive Value for the ARCHITECT High Sensitive Troponin I was evaluated using K2 EDTA tube type for 3 collection time points. The results were calculated using the overall 99th percentile cutoff 26.2 pg/mL).
- Negative Predictive Value in Lithium Heparin Separator: Negative Predictive Value for the ARCHITECT High Sensitive Troponin I was evaluated using Lithium Heparin tube type for 3 collection time points. The results were calculated using the overall 99th percentile cutoff 26.2 pg/mL).
- Negative Predictive Value in Serum Separator: Negative Predictive Value for the ARCHITECT High Sensitive Troponin I was evaluated using Serum tube type for 3 collection time points. The results were calculated using the overall 99th percentile cutoff 26.2 pg/mL).
Arm/Group | Negative Predictive Value in K2 EDTA | Negative Predictive Value in Lithium Heparin Separator | Negative Predictive Value in Serum Separator
Number analyzed (Participants) | 1066 | 1088 | 1029
%nonMI,TnI</=cutoff vs all TnI</=cutoff
  % NPV: 0-2 hours | 98.10 [96.82 to 98.95] | 98.08 [96.81 to 98.95] | 98.73 [97.61 to 99.42]
  % NPV: 2-4 hours | 99.19 [98.25 to 99.70] | 99.05 [98.05 to 99.62] | 99.20 [98.27 to 99.71]
  % NPV: 4-9 hours | 99.23 [98.22 to 99.75] | 99.24 [98.22 to 99.75] | 99.25 [98.26 to 99.76]
Statistical Analysis 1: Comparison: Negative Predictive Value in K2 EDTA; Time point: 0-2 hours; Test type: Superiority or Other; Negative Predictive Value = 98.10, 95% CI 2-sided [96.82 to 98.95]
Statistical Analysis 2: Comparison: Negative Predictive Value in K2 EDTA; Time point: 2-4 hours; Test type: Superiority or Other; Negative Predictive Value = 99.19, 95% CI 2-sided [98.25 to 99.70]
Statistical Analysis 3: Comparison: Negative Predictive Value in K2 EDTA; Time point: 4-9 hours; Test type: Superiority or Other; Negative Predictive Value = 99.23, 95% CI 2-sided [98.22 to 99.75]
Statistical Analysis 4: Comparison: Negative Predictive Value in Lithium Heparin Separator; Time point: 0-2 hours; Test type: Superiority or Other; Negative Predictive Value = 98.08, 95% CI 2-sided [96.81 to 98.95]
Statistical Analysis 5: Comparison: Negative Predictive Value in Lithium Heparin Separator; Time point: 2-4 hours; Test type: Superiority or Other; Negative Predictive Value = 99.05, 95% CI 2-sided [98.05 to 99.62]
Statistical Analysis 6: Comparison: Negative Predictive Value in Lithium Heparin Separator; Time point: 4-9 hours; Test type: Superiority or Other; Negative Predictive Value = 99.24, 95% CI 2-sided [98.22 to 99.75]
Statistical Analysis 7: Comparison: Negative Predictive Value in Serum Separator; Time point: 0-2 hours; Test type: Superiority or Other; Negative Predictive Value = 98.73, 95% CI 2-sided [97.61 to 99.42]
Statistical Analysis 8: Comparison: Negative Predictive Value in Serum Separator; Time point: 2-4 hours; Test type: Superiority or Other; Negative Predictive Value = 99.20, 95% CI 2-sided [98.27 to 99.71]
Statistical Analysis 9: Comparison: Negative Predictive Value in Serum Separator; Time point: 4-9 hours; Test type: Superiority or Other; Negative Predictive Value = 99.25, 95% CI 2-sided [98.26 to 99.76]

6. Primary Outcome: Clinical Performance- Positive Predictive Value (PPV)
Description: The ARCHITECT STAT High Sensitive Troponin-I assay clinical performance was evaluated by calculating the Positive Predictive Value. The ARCHITECT STAT High Sensitive Troponin-I assay results were generated from subject's specimens collected at three collection time points in three tube types (K2 EDTA, Lithium Heparin Separator and Serum Separator).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: %MI,TnI >cutoff vs all TnI > cutoff
Groups:
- Positive Predictive Value in K2 EDTA: Positive Predictive Value for the ARCHITECT High Sensitive Troponin I was evaluated using K2 EDTA tube type for 3 collection time points. The results were calculated using the overall 99th percentile cutoff (26.2 pg/mL).
- Positive Predictive Value in Lithium Heparin Separator: Positive Predictive Value for the ARCHITECT High Sensitive Troponin I was evaluated using Lithium Heparin tube type for 3 collection time points. The results were calculated using the overall 99th percentile cutoff (26.2 pg/mL).
- Positive Predictive Value in Serum Separator: Positive Predictive Value for the ARCHITECT High Sensitive Troponin I was evaluated using Serum tube type for 3 collection time points. The results were calculated using the overall 99th percentile cutoff (26.2 pg/mL).
Arm/Group | Positive Predictive Value in K2 EDTA | Positive Predictive Value in Lithium Heparin Separator | Positive Predictive Value in Serum Separator
Number analyzed (Participants) | 1066 | 1088 | 1029
%MI,TnI >cutoff vs all TnI > cutoff
  % PPV: 0-2 hours | 38.78 [31.92 to 45.98] | 36.82 [30.43 to 43.56] | 35.84 [28.70 to 43.47]
  % PPV: 2-4 hours | 35.68 [29.03 to 42.76] | 35.75 [29.43 to 42.45] | 35.94 [29.16 to 43.16]
  % PPV: 4-9 hours | 36.49 [29.99 to 43.38] | 37.75 [31.71 to 44.09] | 35.05 [28.36 to 42.21]
Statistical Analysis 1: Comparison: Positive Predictive Value in K2 EDTA; Time point: 0-2 hours; Test type: Superiority or Other; Positive Predictive Value = 38.78, 95% CI 2-sided [31.92 to 45.98]
Statistical Analysis 2: Comparison: Positive Predictive Value in K2 EDTA; Time point: 2-4 hours; Test type: Superiority or Other; Positive Predictive Value = 35.68, 95% CI 2-sided [29.03 to 42.76]
Statistical Analysis 3: Comparison: Positive Predictive Value in K2 EDTA; Time point: 4-9 hours; Test type: Superiority or Other; Positive Predictive Value = 36.49, 95% CI 2-sided [29.99 to 43.38]
Statistical Analysis 4: Comparison: Positive Predictive Value in Lithium Heparin Separator; Time point: 0-2 hours; Test type: Superiority or Other; Positive Predictive Value = 36.82, 95% CI 2-sided [30.43 to 43.56]
Statistical Analysis 5: Comparison: Positive Predictive Value in Lithium Heparin Separator; Time point: 2-4 hours; Test type: Superiority or Other; Positive Predictive Value = 35.75, 95% CI 2-sided [29.43 to 42.45]
Statistical Analysis 6: Comparison: Positive Predictive Value in Lithium Heparin Separator; Time point: 4-9 hours; Test type: Superiority or Other; Positive Predictive Value = 37.75, 95% CI 2-sided [31.71 to 44.09]
Statistical Analysis 7: Comparison: Positive Predictive Value in Serum Separator; Time point: 0-2 hours; Test type: Superiority or Other; Positive Predictive Value = 35.84, 95% CI 2-sided [28.70 to 43.47]
Statistical Analysis 8: Comparison: Positive Predictive Value in Serum Separator; Time point: 2-4 hours; Test type: Superiority or Other; Positive Predictive Value = 35.94, 95% CI 2-sided [29.16 to 43.16]
Statistical Analysis 9: Comparison: Positive Predictive Value in Serum Separator; Time point: 4-9 hours; Test type: Superiority or Other; Positive Predictive Value = 35.05, 95% CI 2-sided [28.36 to 42.21]

ADVERSE EVENTS:
Time Frame: Duration of subject emergency department visit: 24 hours.
Groups:
- ARCHITECT STAT High Sensitive Troponin I Assay Testing: All subjects will have their blood tested by the investigational Troponin I assay.
  ARCHITECT STAT High Sensitive Troponin I Assay: Test blood samples from the ARCHITECT STAT High Sensitive Troponin I Assay.
  Results obtained will be used to assess the prognosis of subjects with a troponin result for risk of ACM/MACE in the time frames (30 days and 90 days) after the Emergency Department visit.
  Troponin results will be compared to documented ACM/MACE events at the 30 day and 90 day time points after Emergency Department visit.
Arm/Group | ARCHITECT STAT High Sensitive Troponin I Assay Testing
Serious Adverse Events (participants affected / at risk) | 0/1101
Other Adverse Events (participants affected / at risk) | 0/1101

LIMITATIONS AND CAVEATS:
Some tube types and some time points may not have been obtained for each subject. Every attempt was made to collect all tube types within the time point windows described.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days